CLINICAL TRIAL: NCT04454736
Title: Psychological and Biological Responses to Choral Singing in Mentally Ill, Socially Underprivileged and Privileged Healthy Children and Adolescents: An Open, Single-Arm, Controlled Study
Brief Title: Psychobiological Responses to Choral Singing in Mentally Ill and Healthy Children and Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salzburg (Other)
Collaborators: Universität Mozartuem Salzburg (Unknown); Salzburger Landeskliniken (Other); Paracelsus Medical University (Other); University of Vienna (Other)
Responsible Party: Principal Investigator, Katarzyna Grebosz-Haring, Senior Scientist, Principal Investigator, University of Salzburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Grebosz-Haring SingingStudy
Record Dates: First submitted 2020-02-25; First posted 2020-07-01 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Stress
Keywords: Mental health; Youth; Singing; Music; Stress; Cortisol; Alpha Amylase; Immunoglobulin A
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SBGmentdis (Experimental): Children and adolescents with mental disorders at the Department of Child and Adolescents Psychiatry in Salzburg, Austria
  Interventions: Behavioral: "Amateur" Group Singing
- SBGhealthy (Experimental): Healthy children and adolescents from schools in Salzburg, Austria
  Interventions: Behavioral: "Amateur" Group Singing
- VIEhealthy (Experimental): Members from the Vienna Boys Choir, Austria
  Interventions: Behavioral: "Professional" Group Singing

INTERVENTIONS:
Behavioral: "Amateur" Group Singing — 45-minute singing session led by a professional choirmaster without a therapeutic background once a week
  Arms: SBGhealthy; SBGmentdis
Behavioral: "Professional" Group Singing — 120-minute singing session led by a professional choirmaster without a therapeutic background three times a week. Assessments take place twice a week.
  Arms: VIEhealthy

SUMMARY:
Interventional, three-armed, open, monocentric, medium-term follow-up, pre-test-post-test design, controlled, parallel group study to investigate the effects of a group singing intervention on neuroendocrine (hair cortisol, salivary cortisol, salivary alpha amylase), immune (salivary immunoglobulin A/s-IgA), and psychological (psychological stress, mood, social contacts, emotional and social competence, self-esteem, and quality of life) responses in mentally ill and healthy children and adolescents (N=135, age range 10 -18).

Additionally, the child and adolescent psychiatry group (age range 13-18) takes part in three hour creative workshops every two weeks.

DETAILED DESCRIPTION:
Background: Biopsychological responses to music-related activities (MRA) were examined in various naturalistic settings in adults. Group singing in particular seems to be associated with positive biopsychological outcomes. There is also an emerging view that MRA may play an important role for youth with mental disorders. However, longitudinal research on biopsychological responses to MRA in different clinical and healthy populations among children and adolescents is lacking.

Method: Children and adolescents (age range 10-18) under psychiatric treatment at the Department of Child and Adolescents Psychiatry in Salzburg (n=45), healthy children and adolescents from a school in Salzburg (n=45), and members from the Vienna Boys Choir (n=45) in Austria will be recruited to take part in the study. Subjective measures (mood, stress experience) will be taken pre- and post singing sessions once a week throughout six months. Additionally, salivary biomarkers (cortisol, alpha amylase and IgA), social contacts, and quality of life are assessed. Emotional competence, social competence, self-esteem, and chronic stress levels are measured at the beginning, after three months, at the end, and in a follow-up of the study.

The group of child and adolescent psychiatry taking part in the creative workshops will be additionally assessed via questionnaires regarding emotional regulation, self-esteem, and art experience before and after every workshop. Furthermore, some individuals of the child and adolescent psychiatry group will undergo fMRI evaluation of the brain before and after completion of all creative interventions.

Conclusion: Singing and other creative activities are suggested to benefit mental and physical health in children and adolescents. However, despite the current knowledge, the researchers must better understand the biopsychological mechanisms underlying choral singing in order to determine its full potential, particularly for vulnerable populations. This is the first study to investigate this issue in this population.

ELIGIBILITY:
Inclusion Criteria (Clinical N):

* Written consent to study participation;
* Gender: male, female, different;
* Age: children and adolescents aged ≥ 10 and ≤ 18 years;
* Diagnosis of a psychiatric disorder according to ICD-10;
* Patients are admitted regardless of medication status and are allowed to the medication will continue to be used during the study;
* Additional therapies and medication are recorded and are not an exclusion criterion;
* Musical skills or a certain musical background are not required

Inclusion Criteria (Healthy N):

* Written consent to study participation;
* Gender: male, female, different;
* Age: children and adolescents aged ≥ 10 and ≤ 18 years;
* Musical skills or a certain musical background are not required

Exclusion Criteria (Clinical N):

* Age: children and adolescents aged <10 years and > 18 years;
* Criteria that prevent an application: hearing loss, states of confusion, inability to verbalize;
* Patients with acute externalizing behavior or self-harm/suicidality;
* Existing alcohol addiction or abuse of illegal drugs;

Exclusion Criteria (Healthy N):

* Age: children and adolescents aged <10 years and > 18 years
* Criteria that prevent an application: hearing loss, states of confusion, inability to verbalize

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 135 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change Short-Term Neuroendocrine Stress (Hypothalamic-Pituitary-Adrenal Axis) from pre- to post singing session over six months | every two weeks pre- and post singing sessions for six months
  Biological Stress Marker: Salivary Cortisol
Change Short-Term Immune Function from pre- to post singing session over six months | every two weeks pre- and post singing sessions for six months
  Biological Marker: Salivary Immunoglobulin A
Change from Baseline Chronic Neuroendocrine Stress (Hypothalamic-Pituitary-Adrenal Axis) at three and six months | at the beginning of the study, after three months, at the end of the study after six months, at a follow-up after three months, at a follow up after six months
  Biological Stress Marker: Hair Cortisol
Change Short-Term Neuroendocrine Stress (Autonomic Nervous System) from pre- to post singing session over six months | every two weeks pre- and post singing sessions for six months
  Salivary Alpha-Amylase

SECONDARY OUTCOMES:
Psychological Stress | at the beginning of the study, after three months, at the end of the study after six months, at a follow-up after three months, at a follow up after six months
  Stress and Coping Questionnaire for Children and Adolescents (SSKJ 3-8 R; Lohaus, Eschenbeck, Kohlmann, & Klein-Heßling, 2018)
Mood | every week pre- and post singing sessions for six months
  Multidimensional Mood State Questionnaire (MDBF, short version; Steyer, Notz, Schwenkmezger, & Eid, 1997)
Emotional Skills | at the beginning of the study, after three months, at the end of the study after six months, at a follow-up after three months, at a follow up after six months
  Emotional Competence Questionnaire (EKF; Rindermann, 2009)
Self-Esteem | at the beginning of the study, after three months, at the end of the study after six months, at a follow-up after three months, at a follow up after six months
  Selbstwertinventar für Kinder und Jugendliche (SEKJ; Schöne & Stiensmeier-Pelster, 2016)
Life Quality | once a month for six months
  Pediatric Quality of Life Inventory (PEDsQL; Varni, 2001)
Performance Anxiety | once at the beginning of the study, once after 6 months
  Das State-Trait-Angstinventar (STAI-T adapted; Laux, Glanzmann, Schaffner, & Spielberger 1981)
Social Skills | at the beginning of the study, after three months, at the end of the study after six months, at a follow-up after three months, at a follow up after six months
  Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997)
Evaluation of the choir session | every week post singing sessions for six months
  Liking of the session, liking of the songs, familiarity with the songs (5-point Likert scale; Higher scores mean a better outcome)
Chronical Stress | at the beginning of the study, after three months, at the end of the study after six months, at a follow-up after three months, at a follow up after six months
  Fragebogen zu chronischem Stress im Kindesalter (CSiK; Richartz, Hoffmann, & Sallen, 2009)
Stress Perception | every week pre- and post singing sessions for six months
  Visual Analogue Scale (VAS; 0-100; higher score means a worse outcome)
Prosocial Behavior | every two weeks post singing sessions for six months
  Social Network Map (Tracey & Whittaker, 1990)
Psychological Stability (parents view) | at the beginning of the study, after three months, at the end of the study after six months, at a follow-up after three months, at a follow up after six months
  Child Behavior Checklist (CBCL; Achenbach & Arbeitsgruppe Deutsche Child Behavior Checklist, 1994)
Psychological Stability (children view) | at the beginning of the study, after three months, at the end of the study after six months, at a follow-up after three months, at a follow up after six months
  Youth Self-Report (YSR; Achenbach & Arbeitsgruppe Deutsche Child Behavior Checklist, 1994)
Emotional Control | at the beginning of the study, after three months, at the end of the study after six months, at a follow-up after three months, at a follow up after six months
  Fragebogen zur Erhebung der Emotionsregulation bei Kindern und Jugendlichen (FEEL-KJ; Grob & Smolenski, 2005)
Specific personality and character traits such as curiosity, reward dependency, cooperativity, and self-steering ability | At the beginning of creative workshops, and at a follow-up after three months in the group of children and adolescents with psychiatric disorders
  JTCI Junior Temperament and Character Inventory in Children and Adolescents Psychiatry Group Questionnaire
Current emotional state | Pre and post every creative workshop in the group of children and adolescents with psychiatric disorders
  Positive and negative affect schedule (PANAS)

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Grebosz-Haring, Dr., Principal Investigator — University Mozarteum Salzburg, University of Salzburg; Leonhard Thun-Hohenstein, Prof. Dr., Principal Investigator — Salzburger Landeskliniken Betriebsges.m.b.H.
Locations (3):
- Austria (3):
  - Salzburger Landeskliniken, Universitätsklinik für Kinder- und Jugendpsychiatrie, Salzburg
  - University Mozarteum Salzburg/University of Salzburg, Salzburg
  - University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: July 2020-until the end of the study

REFERENCES:
- [Background] Grebosz-Haring K, Thun-Hohenstein L. Effects of group singing versus group music listening on hospitalized children and adolescents with mental disorders: A pilot study. Heliyon. 2018 Dec 17;4(12):e01014. doi: 10.1016/j.heliyon.2018.e01014. eCollection 2018 Dec. PMID 30582039
- [Background] Grebosz-Haring, K., Thun-Hohenstein, L. (2020). Singing for Health and Wellbeing in Children and Adolescents with Mental Disorders. In R. Heydon, D. Fancourt, A. Cohen (Eds.), The Routledge Companion to Interdisciplinary Studies in Singing: Vol 3 Wellbeing. London: Routledge.
- [Background] Linnemann, A., Schnersch, A., Nater, U. M. (2017). Testing the beneficial effects of singing in a choir on mood and stress in a longitudinal study: The role of social contacts. Musicae Scientiae, 21(2), 195-212.
- [Background] Ali N, Nater UM. Salivary Alpha-Amylase as a Biomarker of Stress in Behavioral Medicine. Int J Behav Med. 2020 Jun;27(3):337-342. doi: 10.1007/s12529-019-09843-x. PMID 31900867